CLINICAL TRIAL: NCT06869213
Title: A Single-arm, Open, Single-center Exploratory Study of Adebrelimab (SHR-1316) in Combination With Chemotherapy for the Perioperative Treatment of Locally Advanced Resectable Esophageal Squamous Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024KT157
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Cancer (EsC)
MeSH Terms: conditions — Esophageal Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab (SHR-1316)+chemotherapy (Experimental)
  Interventions: Drug: Adebrelimab (SHR-1316) + Nab-paclitaxel + Cisplatin

INTERVENTIONS:
Drug: Adebrelimab (SHR-1316) + Nab-paclitaxel + Cisplatin — All subjects were given 3 cycles of neoadjuvant therapy with adebrelimab (1200 mg D1, IV, Q3W)+Nab-paclitaxel(250 mg/m2 D1，IV，Q3W)+Cisplatin(75 mg/m2 D1，IV，Q3W) preoperatively. Within 4-8 weeks of completion of neoadjuvant therapy, all subjects who were suitable for surgery underwent radical surgery, and patients who underwent radical esophageal cancer with R0 resection were given adebrelimab monotherapy postoperatively until disease recurrence or metastasis, toxicity intolerance, initiation of a new antitumor therapy, subject-initiated request to withdraw from the study, and subject's judgement that the subject needed to be withdrawn from the study. The maximum duration of adebrelimab in the adjuvant phase is 16 cycles.

SUMMARY:
This study is a prospective, observational clinical study. In this study, 30 patients with resectable locally advanced esophageal squamous carcinoma will be prospectively enrolled and treated with adebrelimab (SHR-1316) combined with nab-paclitaxel and cisplatin preoperatively and adebrelimab (SHR-1316) single-agent adjuvant therapy postoperatively, to observe the efficacy and safety of this treatment modality, and to provide clinical evidence for the use of PD-L1 monoclonal antibody in perioperative treatment of esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old, regardless of gender；
2. Surgically resectable locally advanced squamous cell carcinoma of the esophagus confirmed by histology or cytology (pre-treatment clinical stage cT1b-cT2, N+ or cT3-cT4a, ANY N according to the 8th edition of AJCC staging);
3. Presence of measurable and/or non-measurable lesions as defined by the criteria for evaluating the efficacy of solid tumors (RECIST v1.1);
4. No prior antitumor therapy for esophageal cancer, including chemotherapy, radiotherapy (including planned radiotherapy during the study period), hormone therapy, and immunotherapy;
5. ECOG PS 0 to 1 point;
6. No contraindication to surgery as evaluated by various organ function tests;
7. Prior to treatment, the following laboratory tests to confirm that bone marrow, liver and kidney function meet the requirements for participation in the study (requiring no blood transfusion or use of hematopoietic stimulating factors (including G-CSF, GM-CSF , EPO, and TPO, etc.) within 14 days prior to screening):

   * Hemoglobin ≥ 90 g/L;
   * White blood cell count ≥ lower limit of laboratory normal;
   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
   * Platelet count ≥100×109/L;
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN);
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN;
   * Prothrombin time ≤ 16 seconds and International Normalized Ratio (INR) ≤ 1.5 x ULN;
   * Creatinine ≤ 1.5 x ULN and Cr clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula);
8. Must understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. malignant tumors other than esophageal cancer within 5 years prior to enrollment (cured limited tumors are not excluded, including cervical carcinoma in situ, basal cell carcinoma of the skin, and carcinoma in situ of the prostate gland; patients with prostate cancer who received hormone therapy and obtained DFS for more than 5 years are not excluded)；
2. Comorbid serious cardiac and cerebrovascular diseases:

   * Congestive heart failure, unstable angina, myocardial infarction, poorly controlled arrhythmia, or cerebrovascular accident of New York Heart Association (NYHA) class II or higher within 12 months prior to enrollment.
   * Medication-uncontrolled hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg) (based on the average of ≥2 measurements)
   * Previous hypertensive crisis or hypertensive encephalopathy
3. Prior history of interstitial lung disease or pneumonia requiring steroid therapy at enrollment；
4. Have a blood-borne infectious disease, including, but not limited to, hepatitis B virus carrier, hepatitis C, syphilis, or HIV;
5. Previous severe allergy to chemotherapeutic agents (paclitaxel or carboplatin) or to any of the monoclonal antibodies;
6. Active autoimmune disease requiring systemic therapy (i.e., immunomodulatory drugs, corticosteroid drugs, or immunosuppressive drugs) within the past 2 years; however, alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered systemic and are permitted and enrollment is allowed;
7. Women during pregnancy;
8. Patients who, in the opinion of the investigator, are not suitable for participation in this study, based on a comprehensive assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR) | Three weeks after surgery of last enrolled subject. Estimate up to 2 years
  The rate of pathologic complete response rate after neoadjuvant therapy
Adverse Events (AE) | about 2 years
  Incidence and grade (including serious adverse events and immunization-related adverse events), as determined by NCI-CTCAE 5.0 criteria

SECONDARY OUTCOMES:
R0 resection rate | Three weeks after surgery of last enrolled subject. Estimate up to 2 years
  The R0 resection rate of esophagectomy
Major pathologic response rate | Three weeks after surgery of last enrolled subject. Estimate up to 2 years.
  The percentage of subjects with ≤10% survival tumor cells in the resected specimens after neoadjuvant therapy accounted for all subjects who received surgical treatment.
Objective Response Rate | Estimate up to 2 years
  The percentage of patients having a complete response or a partial response to protocol treatment. Objective response will be measured by RECIST 1.1.
Event-free survival (EFS) | Estimate up to 2 years
  The length of time between signing the informed consent form and the occurrence of any of the following events: disease progression, disease recurrence, or death from any cause
1-year event-free survival rate (1-year EFS) | Estimate up to 2 years
  The percentage of subjects who were free of the occurrence of any of the events(disease progression, disease recurrence, or death from any cause) from the start of study enrolment to 12 months later.
Disease-free survival (DFS) | about 2 years
  The time from enrolment (ICF signing) to disease recurrence or death due to disease progression.
1-year disease-free survival rate (1-year DFS) | about 2 years
  The percentage of subjects who were free of disease recurrence or death from the start of study enrolment to 12 months later.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, China